CLINICAL TRIAL: NCT00105742
Title: Audiology Visits After Screening for Hearing Loss: An RCT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IIR 99-377
Record Dates: First submitted 2005-03-16; First posted 2005-03-17 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2006-07

CONDITIONS: Hard of Hearing
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Procedure: Diagnosis

INTERVENTIONS:
Procedure: Diagnosis

SUMMARY:
Hearing impairment is one of the most common disabilities in veterans. The decreased ability to communicate is troubling in itself, but the strong association of hearing loss with functional decline and depression adds further to the burden on the hearing-impaired. Although hearing amplification improves quality of life, hearing evaluations are offered infrequently to older patients. Only 25 percent of patients with aidable hearing loss receive treatment. Up to 30 percent of patients who receive hearing aids do not use them. We contend that an effective formal screening program should identify hearing-impaired patients who are motivated to seek evaluation and who derive benefit from treatment.

DETAILED DESCRIPTION:
Background:

Hearing impairment is one of the most common disabilities in veterans. The decreased ability to communicate is troubling in itself, but the strong association of hearing loss with functional decline and depression adds further to the burden on the hearing-impaired. Although hearing amplification improves quality of life, hearing evaluations are offered infrequently to older patients. Only 25 percent of patients with aidable hearing loss receive treatment. Up to 30 percent of patients who receive hearing aids do not use them. We contend that an effective formal screening program should identify hearing-impaired patients who are motivated to seek evaluation and who derive benefit from treatment.

Objectives:

The first specific aim is to determine if formal screening programs for hearing loss can increase visits to audiologists. The second specific aim is to determine which specific screening strategy leads to the most frequent audiology visits.

Methods:

Our four-armed randomized clinical trial compares three screening strategies (physiologic testing, a self-report questionnaire, and combined use of both physiologic and self-report testing), against a control arm (usual care). Physiologic testing was done with the Audioscope, a portable otoscope that emits tones from selected frequencies at a variety of loudness levels. The self-report questionnaire was the screening version of the Hearing Handicap Inventory of the Elderly questionnaire (HHIE-S), which quantifies the social and emotional handicap from hearing loss. Patients aged 50 and older who did not wear hearing aids were recruited from the outpatient clinics at the VA Puget Sound Health Care System. Only patients who were eligible for VA-issued hearing aids were enrolled in this trial. Patients randomized to the control arm were not screened. Patients screened with both the Audioscope and HHIE-S were referred to the audiology service for evaluation if either of the tests was positive. All patients, regardless of screening status, were followed to determine how many patients in each arm subsequently visit an audiologist.

The primary outcome is the percentage of patients who contact the audiology service within 6 months of the date of screening. Secondary outcomes include: 1) the number of cases of hearing loss detected; 2) the number of dispensed hearing aids; 3) self-rated communication ability; 4) hearing-related quality of life; and 5) rates of hearing aid adherence. Costs of screening and subsequent treatment were collected. The study is not powered to determine cost-effectiveness, but to pilot calculations of the costs to implement the screening program will be made. An intention-to-screen analysis will be used to minimize bias due to subject self-selection.

Status:

Enrollment and follow-up is complete. Outcomes data are currently being analyzed.

ELIGIBILITY:
Inclusion Criteria:

Hearing impaired

Exclusion Criteria:

Not Hearing Impaired

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1400 (Estimated)
Dates: Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
Better diagnois of hearing problems

SECONDARY OUTCOMES:
Improved quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Bevan Yueh, MD MPH, Principal Investigator — VA Puget Sound Health Care System Seattle Division, Seattle, WA
Locations (1):
- VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington, United States

REFERENCES:
- [Result] Collins MP, Souza PE, Yueh B. Effects of group versus individual hearing aid visits. Journal of The American Auditory Society. 2007 Mar 1; 31(1):34.
- [Result] Yueh B, Collins MP, Souza PE. Effects of depression on self-report hearing outcomes. Journal of The American Auditory Society. 2007 Mar 1; 32(1):32.
- [Result] Yueh B, Collins MP, Souza PE, Heagerty PJ, Liu CF, Boyko EJ, Loovis CF, Fausti SA, Hedrick SC. Screening for Auditory Impairment-Which Hearing Assessment Test (SAI-WHAT): RCT design and baseline characteristics. Contemp Clin Trials. 2007 May;28(3):303-15. doi: 10.1016/j.cct.2006.08.008. Epub 2006 Aug 30. PMID 17030153
- [Result] Yueh B, Collins MP, Souza PE, Boyko EJ, Loovis CF, Heagerty PJ, Liu CF, Hedrick SC. Long-term effectiveness of screening for hearing loss: the screening for auditory impairment--which hearing assessment test (SAI-WHAT) randomized trial. J Am Geriatr Soc. 2010 Mar;58(3):427-34. doi: 10.1111/j.1532-5415.2010.02738.x. PMID 20398111
- [Result] Yueh B, Shapiro N, MacLean CH, Shekelle PG. Screening and management of adult hearing loss in primary care: scientific review. JAMA. 2003 Apr 16;289(15):1976-85. doi: 10.1001/jama.289.15.1976. PMID 12697801
- [Result] Bogardus ST Jr, Yueh B, Shekelle PG. Screening and management of adult hearing loss in primary care: clinical applications. JAMA. 2003 Apr 16;289(15):1986-90. doi: 10.1001/jama.289.15.1986. PMID 12697802
- [Result] Yueh B. Digital hearing aids. Arch Otolaryngol Head Neck Surg. 2000 Nov;126(11):1394-7. doi: 10.1001/archotol.126.11.1394. No abstract available. PMID 11074842
- [Result] Kezirian EJ, White KR, Yueh B, Sullivan SD. Cost and cost-effectiveness of universal screening for hearing loss in newborns. Otolaryngol Head Neck Surg. 2001 Apr;124(4):359-67. doi: 10.1067/mhn.2001.113945. PMID 11283492
- [Result] Yueh B, Souza PE, McDowell JA, Collins MP, Loovis CF, Hedrick SC, Ramsey SD, Deyo RA. Randomized trial of amplification strategies. Arch Otolaryngol Head Neck Surg. 2001 Oct;127(10):1197-204. doi: 10.1001/archotol.127.10.1197. PMID 11587599